CLINICAL TRIAL: NCT02508038
Title: TCR-αβ+ and CD19+ Depleted KIR/KIR Ligand-mismatched Haploidentical Hematopoietic Stem Cell Transplant and Zoledronate for Pediatric Relapsed/Refractory Hematologic Malignancies and High Risk Solid Tumors
Brief Title: Alpha/Beta CD19+ Depleted Haploidentical Transplantation + Zometa for Pediatric Hematologic Malignancies and Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW13090; NCI-2015-01163 (Registry Identifier: NCI Trial ID); 2015-0290 (Other: Institutional Review Board); A536700 (Other: UW Madison); SMPH\PEDIATRICS\PEDIATRICS (Other: UW Madison); Protocol Version 10/12/2021 (Other: UW Madison)
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Myelodysplastic Syndrome; Myeloproliferative Syndrome; Rhabdomyosarcoma; Ewing Sarcoma; Primitive Neuroectodermal Tumor; Osteosarcoma; Neuroblastoma
Keywords: alpha beta depleted; alphabeta; TCR alpha beta depleted; alpha beta; haploidentical; Zoledronate; Zoledronic acid; Pediatric cancers; alfa beta; αβ T cell depleted HSCT; alpha beta T cell and B cell depleted HSCT; haploidentical HSCT
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Rhabdomyosarcoma; Sarcoma, Ewing; Neuroectodermal Tumors, Primitive; Osteosarcoma; Neuroblastoma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TCRαβ+/CD19+ depleted Haploidentical HSCT+ Zoledronate (Experimental): Patients with high-risk leukemia (who are at least one year of age and who have not received TBI as conditioning for a previous HSCT) will receive myeloablative conditioning with ATG, Fludarabine, Thiotepa, and TBI. All other subjects will undergo a reduced-intensity conditioning regimen consisting of ATG, Fludarabine, Thiotepa, and Melphalan prior to transplant with a KIR/KIR ligand mismatched haploidentical donor peripheral blood stem cell graft depleted of TCR-αβ+ and CD19+ cells. Patients will receive 5 doses of zoledronate (at 28 day intervals) starting 28 days after stem cell transplant.
  Interventions: Procedure: TCRαβ+/CD19+ depleted Haploidentical HSCT; Drug: Zoledronate

INTERVENTIONS:
Procedure: TCRαβ+/CD19+ depleted Haploidentical HSCT — Patients with high-risk leukemia will receive myeloablative conditioning. All other patients will undergo a reduced-intensity conditioning with ATG, Fludarabine, Thiotepa and Melphalan followed by transplant with a KIR/KIR (Killer cell immunoglobulin-like recetptor) ligand mismatched haploidentical donor peripheral blood stem cell graft depleted of TCRab+ cells and CD19+ cells using the CliniMACS System.
Drug: Zoledronate — Given IV. Patients will receive five doses of Zoledronate (each 1.25 mg/m2 at a 28 day interval) following transplant.
  Other Names: Zoledronic Acid; Zometa

SUMMARY:
This phase I trial studies the safety of transplantation with a haploidentical donor peripheral blood stem cell graft depleted of TCRαβ+ cells and CD19+ cells in conjunction with the immunomodulating drug, Zoledronate, given in the post-transplant period to treat pediatric patients with relapsed or refractory hematologic malignancies or high risk solid tumors.

DETAILED DESCRIPTION:
CONDITIONING REGIMENS: Patients with high-risk leukemia will receive myeloablative conditioning with anti-thymocyte globulin intravenously (IV) over 4-6 hours on days -12 through -9, Fludarabine IV over 30 minutes on days -8 through -5, Thiotepa IV every every 12 hours on day -4 and Total Body Irradiation (TBI) on days -3 through -1. All other patients receive reduced intensity conditioning consisting of anti-thymocyte globulin intravenously (IV) over 4-6 hours on days -12 through -9, fludarabine IV over 30 minutes on days -8 through -5, thiotepa IV over 4 hours every 12 hours on day -4, and melphalan IV on days -3 and -2.

PERIPHERAL BLOOD STEM CELL TRANSPLANTATION: Patients undergo TCR-alpha/beta+ and CD19+ depleted KIR/KIR ligand-mismatched haploidentical donor peripheral blood stem cell transplantation on day 0. If the graft contains less than 4 x 10^6 CD34+ cells/kg, a second HSC graft may be administered.

PROPHYLAXIS FOR GVHD: Patients receiving a graft containing > 25 x 10^3 CD3+ TCR alpha/beta+ cells receive mycophenolate mofetil IV twice daily over 2 hours on days 1 to 30 with a rapid taper. Patients with TCR alpha/beta+ cells exceeding 100,000/kg also receive tacrolimus IV continuously or orally (PO) every 12 hours on days 0-90 with a taper at the discretion of the Principal Investigator.

ZOLEDRONATE ADMINISTRATION: Patients will receive five doses of Zoledronate (IV) at 28 day intervals beginning on Day +28 post-HSCT.

Follow-up assessments will occur after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Availability of an eligible haploidentical donor
* Hematologic malignancy or solid tumor
* Patients with more than one malignancy (hematologic or solid tumor) are eligible
* Patients with hematologic malignancy must have no HLA identical sibling or suitable unrelated donor OR time needed to find an acceptable unrelated donor match would likely result in disease progression such that the patient may become ineligible for any type of potentially curative transplant

  * Relapsed or primary therapy-refractory AML with bone marrow blast < 20%
  * High-risk refractory or relapsed ALL in patients for whom transplantation is deemed indicated (relapse occurring < 30 months from diagnosis, patients relapsing after previous allogeneic transplant, relapse after 2nd remission, primary induction failure or hypodiploidy)
  * Relapsed Hodgkin lymphoma unable to achieve 2nd remission or Very Good Partial Response (VGPR) and therefore ineligible to receive autologous hematopoietic stem cell transplant (auto-HSCT)
  * Hodgkin lymphoma relapsing after auto-HSCT
  * Primary refractory or relapsed non-Hodgkin lymphoma unable to achieve 2nd remission or VGPR and therefore ineligible to receive auto-HSCT
  * Non-Hodgkin lymphoma relapsing after auto-HSCT
  * Myelodysplastic Syndrome/Myeloproliferative Syndrome

Solid Tumor

* Patients with solid tumor must have failed or have been ineligible to receive auto-HSCT or if auto-HSCT would not offer > 20% chance of cure
* Neuroblastoma

  * high risk with relapsed or refractory disease
* Soft tissue sarcomas (Rhabdomyosarcoma, Ewing sarcoma, Primitive Neuroectodermal Tumor or other high-risk extracranial solid tumors)

  * Relapsed or primary refractory metastatic
  * 1st complete remission, but very high-risk features (i.e., < 20% survival with conventional therapy)
* Osteosarcoma

  * Failure to achieve Complete Response (CR) following initial therapy
  * Relapsed with pulmonary or bone metastases and did not achieve a CR with surgery and/or chemotherapy
* Karnofsky (patients > 16 years) or Lansky (patients 16 years or older) performance score of ≥ 60
* Life expectancy of ≥ 3 months
* Patient must have fully recovered from acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Study enrollment no earlier than 3 months after preceding HSCT
* Glomerular Filtration Rate (GFR) ≥ 60 ml/min/1.73m2
* Total bilirubin < 3 mg/dL
* ALT (alanine aminotransferase, SCPT) ≤ 5 x Upper LImit of Normal (ULN) for age
* Ejection fraction of > 40% by Multigated Acquisition Scan (MUGA) or echocardiogram
* No evidence of dyspnea at rest
* No supplemental oxygen requirement
* If measured, carbon monoxide diffusion capacity (DLCO) >50%
* No severe peripheral neuropathy, signs of leukoencephalopathy or active Central Nervous System (CNS) infection
* Patients with seizure disorders may be enrolled if seizures are well controlled on anticonvulsant therapy
* If of reproductive potential, negative pregnancy test and willing to use effective birth control method
* Informed consent from patient or legal guardian (if patient is minor)

Inclusion Criteria for Donors:

* Donor must be 18 years of age minimum, 65 years of age maximum
* Donor must be in good general health as determined by evaluating medical provider
* Must meet donor criteria for human cells, tissues, and cellular and tissue-based products per Code of Federal Regulations 21 CFR 1271, subpart C. Specifically:

  * Donor screening in accordance with 1271.75 indicates that the donor:

    * Is free from risk factors for, and clinical evidence of, infection due to relevant communicable disease agents and diseases; and
    * Is free from communicable disease risks associated with xenotransplantation; and
  * The results of donor testing for relevant communicable disease agents in accordance with 1271.80 and 1271.85 are negative or nonreactive, except as provided in 1271.80(d)(1).
* Haploidentical by HLA-typing
* Preference will be given to donors who demonstrate KIR incompatibility with recipient HLA class I ligands defined as the donor expressing a KIR gene for which the corresponding HLA class I ligand is not expressed by the recipient.
* Negative testing for relevant communicable diseases:

  * Hepatitis B surface antigen (HBsAg)
  * Hepatitis B core antibody (Anti-HBc)
  * Hepatitis C antibody (Anti-HCV)
  * HIV 1 & 2 antibody (Anti-HIV-1, 2 plus O)
  * HTLV I/II antibody (Anti-HTLV I/II)
  * RPR (Syphilis TP)
  * CMV (Capture CMV)
  * MPX for: HepB (HBV-PCR), HepC (HCV-PCR), HIV (HIV-PCR)
  * NAT for West Nile Virus (WNV-PCR)
  * T. Cruzi - EIA (Chagas)

Exclusion Criteria:

* Pregnant or breast-feeding
* HIV infection
* Heart failure or uncontrolled cardiac rhythm disturbance
* Uncontrolled, Serious Active Infection
* Prior organ allograft
* Significant serious intercurrent illness unrelated to cancer or its treatment not covered by other exclusion criteria expected to significantly increase the risk of HSCT
* Any mental or physical condition, in the opinion of the PI (or PI designee), which could interfere with the ability of the subject (or the only parent or legal guardian available to care for the subject) to understand or adhere to the requirements of the study
* Enrollment in any other clinical study from screening up to Day 100 (unless PI judges such enrollment would not interfere with endpoints of this study)

Exclusion Criteria for Donors:

* Lactating females
* Pregnant females

Ages: 7 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-02-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute graft versus host disease (GVHD) | Within 100 days post-transplantation
Incidence of graft failure | At day 28

SECONDARY OUTCOMES:
Immune reconstitution | Up to 1 year
  Immune reconstitution outcomes, as determined by immune cell analysis.
Performance of the CliniMACS Reagent System utilizing the CliniMACS TCRαβ-biotin and CliniMACS CD19 reagent to produce a graft with defined cell content. | Day 0
  The performance of the CliniMACS Reagent System will be evaluated by measuring the number of viable stem cells, TCRαβ+ cells, TCRγδ+ cells, NK cells and B cells in the hematopoietic stem cell graft.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Capitini, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/